CLINICAL TRIAL: NCT00379392
Title: Mental Imagery to Reduce Motor Deficits in Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrew Butler, PhD, Prinicipal investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 338-2003; R21AT002138-03 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
Keywords: Stroke; Mental Imagery; Constraint Induced Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mental Imagery and CIT (Experimental): Mental Imagery and Constraint Induced Therapy
  Interventions: Procedure: Mental Imagery and Constraint induced therapy
- Mental Imagery only (Active Comparator): Mental Imagery only
  Interventions: Behavioral: Mental Imagery only

INTERVENTIONS:
Behavioral: Mental Imagery only — Listening to an audio tape to enhance mental imagery of functional activities of the affected upper extremity
  Arms: Mental Imagery only
Procedure: Mental Imagery and Constraint induced therapy — Listening to an audio tape to enhance mental imagery AND participation in constraint induced therapy
  Arms: Mental Imagery and CIT

SUMMARY:
The primary aim of the proposed study is to collect data in an effort to estimate the clinical effectiveness of implementing repetitive task practice (RTP) in addition to mental imagery training (MIT) to improve upper extremity motor function and the quality of life of chronic stroke patients.

DETAILED DESCRIPTION:
Stroke is the leading cause of chronic disability in the United States, and lack of upper limb motor control is a major contributor to stroke-related disability. Physical and occupational therapy treatments are most commonly used to reduce long-term disability. Unfortunately, little scientific evidence exists to best target patients for therapy, define when such therapies should be provided, or even to identify the best therapies themselves. A recent National Institutes of Health consensus panel decided that there were only three therapeutic techniques with supporting scientific evidence, and for only one of these techniques, constraint induced therapy, was there evidence from a randomized trial.

The imagination, probably our most under-utilized health resource, can be used to remember and recreate the past, develop insight into the present, influence physical health, improve creativity and inspiration, and anticipate possible futures. All of us have, to some extent, experienced the effects of the imagination on the body. In recent years, data have suggested that mental practice can improve the performance of motor skill behaviors. These studies have generally shown that healthy volunteers who train with their minds on a specific task usually show better performance compared with a those that did not practice, although less than those who train physically.

To date, only a few small attempts to use mental practice in rehabilitation have been tried. A study in subacute stroke patients comparing the possibility and effectiveness of a program that combined imagery and physical therapy with a program of physical therapy only, showed that combining the two therapies is a clinically feasible, cost-effective addition to therapy that may improve functional outcomes more than participation in physical therapy only. Thus, mental practice in physical rehabilitation offers a potential way to improve motor recovery after damage to the brain.

One approach to improve arm function among patients with stroke is intensive repetitive task practice (RTP). This treatment can take the form of functional training alone or also include other ways encouraged within constraint induced (CI) movement therapy. Repetitive activities often used in physical or occupational therapy may also improve health related quality of life. While intense treatment, such as CI therapy, to overcome arm impairment may prove to be helpful, such therapy is expensive because it relies on one-on-one interaction between the patient and rehabilitation therapist. New therapeutic treatments to help existing therapy that offer helpful and money saving alternatives must be developed to improve arm use, and also, stroke survivors' quality of life.

While RTP and mental imagery may be promising treatments, we do not clearly understand the changes that may occur in the brain's of patients who have had a stroke following any physical rehabilitation. A few studies using positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) measures have shown the blood flow changes in the brain during physical movement following CIT. If the way in which recovery of motor function after stroke were better understood, better decisions could be made regarding the best selection of specific treatment strategies.

The primary aim of the proposed study is to collect data in an effort to estimate the clinical effectiveness of implementing RTP in addition to mental imagery training (MIT) to improve upper extremity motor function and the quality of life of chronic stroke patients. One group in this study will be asked to "mentally rehearse" a series of upper limb functional motor tasks for one and a half hours per day (3-30 minute sessions), with the guidance of an audio tape, for a total of 21 hours over two weeks. Another group will undergo 10 days (6 hours per day) RTP with a licensed rehabilitation specialist as well as listen to the same MIT tape for one and a half hours per day (3-30 minute sessions. Motor function and quality of life will be measured on two occasions: before the intervention and immediately after the intervention. A unique aspect of this study will be to obtain the fMRI data on a subset of patients enrolled in each group. Everything involving this study will be done at the Center for Rehabilitation Medicine at Emory University School of Medicine and at the Emory University Hospital.

This study represents one of the first tries at using mental imagery in addition to a physical rehabilitation for the recovery of movement after stroke and, to our knowledge, the first try to use fMRI to look at changes in the brain after mental training. The results of this study may allow us to learn more about the relationship between rehabilitation and brain function after stroke, as well as confirm the idea that actual changes in the brain are related to improving movement in the body.

This study uses an new therapeutic method along with well accepted methods (RTP) in an effort to improve arm movement of patients who have had a stroke. A thorough approach will be used to determine how the use of mental imagery along with RTP can change movement of the arm and the quality of life of patients who have had a stroke using proven clinical tests to determine movement performance and patients' quality of life. Furthermore, precise brain functioning tests (i.e. fMRI) will be performed to better understand the actual changes that happen in the brain when stroke patients have improved movement in their arm.

Should the use of MIT and RTP be better than RTP or MIT alone, a many year randomized clinical trial would be suggested to determine the helpfulness of using mental imagery training with RTP to improve arm function and the quality of life of patients with stroke. The benefits of this would be reduced costs for arm rehabilitation among certain patients who have had strokes and a better way for rehabilitation centers to prescribe and provide therapy targeting the arm. Because of shorter lengths of stay and fewer number of therapy sessions allowed for in- and out-patient services for stroke survivors, the use of additional and different delivery systems, such as mental imagery, become very important.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum Motor Criteria Active wrist extension of no less than 10 degrees, 10 degrees of thumb abduction/extension and at least two additional digits. Must be able to perform at least 3 times in 1 minute.
2. Passive Range of Motion At least 90 degrees of shoulder flexion and abduction, 45 degrees of shoulder external rotation, no less than -30 degrees of elbow extension, 45 degrees of forearm supination (from neutral), 45 degrees of forearm pronation (from neutral), wrist extension to neutral, finger extension (all digits) such that no MCP joint has greater than a 30 degree contracture.
3. Participants who are 3-12 months post-stroke (first-time clinical CVA) of ischemic or hemorrhagic type at the beginning of the intervention.
4. Participants with sensory loss will be eligible.
5. Participants must score at least 24 on the MMSE. Memory deficits associated with dementia are the main concern with this inclusion criterion.
6. Balance Criteria: Participants must be able to transfer to and from the toilet independently and safely, stand from a sitting position and maintain standing balance independently for at least two minutes with or without their own upper extremity support.
7. Each participant must have physician approval for participation in the therapy to rule out major medical problems.
8. Participants must be over the age of 18 years. No upper age limits will be set.
9. Participants must have sufficient endurance and stamina determined by clinical judgment to carry out the requirements of the CI therapy trial.
10. Participants with unilateral perceptual neglect will be accepted if they meet the other inclusion criteria.
11. Participants on medication will not be excluded. Subjects will be excluded if they have received Botox injections to their affected UE less than 3 months prior to participation, if they have received Phenol block injections less than 12 months prior to participation, if they are receiving intrathecal Baclofen, or if they are receiving Baclofen or Dantrium orally at the time of the study.
12. Transportation to and from Emory Center for Rehabilitation.

Exclusion Criteria:

1. Score of less than 24 on the MMSE.
2. A first stroke less than 3 months or more than 12 months prior to enrollment.
3. Less than 18 years of age.
4. Clinical judgment of excessive frailty or lack of stamina (e.g., cannot attend to instructions, stay awake, engage in functional activities, etc.).
5. Serious uncontrolled medical conditions.
6. Excessive pain in any joint or more affected extremity that could limit ability to cooperate with the intervention, as judged by the examining clinician.
7. Passive ROM less than 90 degrees of shoulder flexion and abduction, less than 45 degrees of shoulder external rotation, greater than 30 degree flexion contracture of elbow, less than 45 degrees of forearm supination and pronation from neutral, less than neutral wrist extension and greater than 30 degree flexion contracture of any MCP joint.
8. Unable to stand independently for 2 minutes, transfer independently to and from the toilet or perform sit-to-stand.
9. Have received injections of anti-spasticity drugs into upper extremity musculature within the past 3 months, or wish to have drugs injected in the foreseeable future.
10. Receiving any anti-spasticity drugs orally at the time of expected participation.
11. Received phenol injections less than 12 months prior to participation.
12. Damage to the parietal area of the brain

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-01; Primary Completion 2008-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Pre-treatment, Post-treatment, and 3 month follow-up
Fugl-Meyer Motor Assessment Test | Pre-treatment, Post-treatment, and 3 month follow-up
Movement Imagery Questionnaire | Pre-treatment, Post-treatment, and 3 month follow-up
Vividness of Movement Imagery Questionnaire | Pre-treatment, Post-treatment, and 3 month follow-up
Center for Epidemiologic Studies Depression scale | Pre-treatment, Post-treatment, and 3 month follow-up
Stroke Impact Scale | Pre-treatment, Post-treatment, and 3 month follow-up

SECONDARY OUTCOMES:
Sirigu's break test | Pre-treatment, Post-treatment, and 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Butler, PhD, MPT, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States